CLINICAL TRIAL: NCT03698643
Title: Impact of New Interventional Imaging Modality Use (Angio-CT) on Patient Radiation Exposure in Transarterial Chemoembolization
Brief Title: Impact of New Interventional Imaging Modality Use on Patient Radiation Exposure in Transarterial Chemoembolization
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0136
Record Dates: First submitted 2018-09-12; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Hepatic Tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Transarterial chemoembolization (TACE) is the most performed endovascular interventional radiology (IR) procedure. TACE procedures are performed in an IR suite, most of which are equipped with floor-based flat-panel robotic C-arm allowing two-dimensional imaging. Cone-beam computed tomography (CBCT) has been developed to allow three-dimensional navigation but has several limitations such as reduced signal to noise ratio and small field-of-view, and seems to have negative impact on patient radiation exposure. Another option to perform 3D imaging is called angio-CT which combines a CT-scan and a floor-based flat-panel robotic C-arm in a single IR suite. Even if some publications have shown benefit of angio-CT in TACE procedures in Japan, no study about angio-CT in liver IR procedures has been conducted in the occidental world so far. The purpose of our study was to assess the impact of angio-CT use on patient radiation exposure and treatment quality in TACE procedures compared to CBCT.

This before-after study consisted of a review of consecutive TACE procedures performed between January 2016 and September 2017 in our institution with two different imaging modalities, defining two study groups (C-arm with CBCT versus angio-CT).

ELIGIBILITY:
Inclusion criteria:

* Age > or = 18 years
* primary or secondary liver tumor(s)
* TACE approved by multidisciplinary tumor meeting

Exclusion criteria:

- TACE not performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TACE sessions performed on adult patients with primary or secondary liver tumor(s) after multidisciplinary tumor meeting approval
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Patient effective radiation dose per TACE | 1 day
  Patient effective radiation dose (mSv) per TACE :
  Dose-area product (in mGy/cm^2) and dose-length product (in mGy/cm) will be combined and converted to report effective dose (in mSv).

SECONDARY OUTCOMES:
Air kerma per TACE | 1 day
  Air kerma (in mGy) per TACE
Fluoroscopy time per TACE | 1 day
  Fluoroscopy time (in sec) per TACE
Number of CBCT acquisitions per TACE | 1 day
  Number of CBCT acquisitions per TACE
Number of CT acquisitions per TACE | 1 day
  Number of CT acquisitions per TACE
Treatment targeting | 1 day
  Assessed on control CBCT or CT and graded into 3 classes : fully targeted, partially targeted or untargeted.
Tumor response | 1 day
  Assessed on follow-up CT or MRI and graded into 3 classes : response, tumor stability or progression.

CONTACTS AND LOCATIONS:
Overall Officials: BORIS GUIU, PU-PH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC